CLINICAL TRIAL: NCT06199544
Title: Effect of Unani Medicine Coded Formulations for the Management of Anomalies Associated With Polycystic Ovarian Syndrome
Brief Title: Effect of Unani Medicine for the Management of Anomalies Associated With Polycystic Ovarian Syndrome
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamdard University (Other)
Responsible Party: Principal Investigator, Leena Hameed, Assistant professor, Hamdard University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HamdardUniversity
Record Dates: First submitted 2023-01-29; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Comparative Study
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Experimental): metformin 500 mg twice a day
  Interventions: Drug: Metformin
- Picolin group (Experimental): Picolin 500mg thrice a day
  Interventions: Drug: Metformin
- Rasoline (Experimental): Rasoline 500mg thrice a day
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Comparing the effect of drugs on symptoms of PCOS
  Other Names: Picolin; Rasoline

SUMMARY:
Currently available medications for PCOS are symptom(s) oriented but have limitations because of its complex pathophysiology. The most preferred drug against PCOS is metformin which act as an insulin sensitizer to improve insulin-glucose metabolism and anovulatory cycles in PCOS. However, its use is associated with various side effects such as bloating, diarrhea and nausea. Thus, it is imperative to explore various other alternatives to combat this gynecological problem.

DETAILED DESCRIPTION:
Polycystic ovarian syndrome (PCOS) is a common endocrine disorder in reproductive age women, with a prevalence between 5%-15%. Currently, sedentary lifestyle, excessive intake of junk food and increasing prevalence of obesity has been associated with rise in the incidence of PCOS.

ELIGIBILITY:
Inclusion criteria No complications record of reproductive system, 4) PCOS diagnosed using Rotterdam criteria fulfilling any two of the following: (i) Menstrual irregularity or oligo-/anovulation, (ii) Hyperandrogenism (clinically and/or biochemically), (iii) Polycystic appearance on ultrasound

Exclusion criteria

1) Patients with severe adverse drug reactions, 2) Record of cardiovascular, diabetes, hepatic and neoplastic disorders or other concurrent medical illnesses, 3) Hormonal contraceptive used within 6 months, or anti-obesity drugs within 3 months of the study, 4) Irregular menstrual bleeding other than PCOS and 5) Positive pregnancy test.

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in the menstrual regularity of the patient | 1 year
  The lengths and duration of menstrual cycle of patients will be measured

CONTACTS AND LOCATIONS:
Locations (1):
- Shifa ul mulk memorial hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No